CLINICAL TRIAL: NCT04117152
Title: Multicenter International Observational Study to Identify Trajectories of Cardiac Allograft Vasculopathy After Heart Transplantation and Their Specific Determinants
Brief Title: Trajectories of Cardiac Allograft Vasculopathy After Heart Transplantation
Acronym: TRAJ-CAV
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); European Georges Pompidou Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ParisTRCOT_CAV
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Heart Transplantation; Allograft Arteriopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Latent class mixed modeling — To identify CAV trajectories after heart transplantation using a contemporary unsupervised trajectory-based approach known as latent class mixed modeling

SUMMARY:
This project aims: i) to identify Cardiac Allograft Vasculopathy (CAV) trajectories after heat transplantation using latent class mixed modeling, ii) to characterize the global and specific determinants of different trajectories and iii) to provide an easily accessible tool to project individual probability of CAV trajectory belonging.

DETAILED DESCRIPTION:
Background:

Cardiac Allograft Vasculopathy (CAV) is the third cause of late mortality and the leading cause of late allograft dysfunction. The field of heart transplantation currently lacks longitudinal description of CAV profiles. Identifying relevant CAV trajectories, or evolution profiles, and their respective determinants is an unmet clinical need. CAV trajectories requires an additional level of understanding and characterization over the current paradigm. Understanding the mechanisms and clinical factors involved in the development of CAV will be useful to provide a more nuanced picture of disease progression, which may ultimately contribute to risk stratification and ultimately guiding the care of HTx patients.

Main Outcome(s) and Measure(s):

* Identification of CAV trajectories after transplantation using an unsupervised latent class mixed modeling. CAV angiograms were recorded per center protocol for all patients after transplantation. CAV was graded according to the current ISHLT classification as CAV 0 (not significant), 1 (mild), 2 (moderate) and 3 (severe).
* Determination of clinical, functional, structural, immunological factors associated with the trajectories. In the derivation cohort, the associations between CAV trajectories and clinical, histological, functional, and immunological parameters at the time of transplantation, during the first year and at one-year post-transplant were assessed using multinomial logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Heart recipient with at least two coronary angiograms after heart transplantation,
* Heart recipient over 18 years of age.

Exclusion Criteria:

* Patient with < 2 coronary angiograms during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart recipients aged over 18 and of all genders recruited between 2004 and 2015 from European and North American centers, who had at least two coronary angiograms during follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Identification of trajectories of Cardiac Allograft Vasculopathy (CAV) | 10 years post-transplant
  Identification of different evolutive profiles of CAV using latent classes mixed models. Each coronary angiogram was graded from 0 (no CAV) to 3 (severe CAV) according to ISHLT classification.

SECONDARY OUTCOMES:
Identification of the specific determinants of CAV trajectories | From transplantation to 1-year post-transplant
  Identification of immune and non-immune determinants using multivariable multinomial logistic regression.
Early prediction of CAV trajectories | 10 years post-transplant
  Probability of belonging to each trajectory according to the baseline angiogram and independent risk factors for CAV
Patients and allograft survival probability according the CAV trajectory | 10 years post-transplant
  Comparison of prognosis according the CAV trajectory

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Principal Investigator — Paris Transplant Group
Locations (3):
- Jon Kobashigawa, Los Angeles, California, United States
- Maarten Naesens, Leuven, Belgium
- Paris Transplant Group, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loupy A, Coutance G, Bonnet G, Van Keer J, Raynaud M, Aubert O, Bories MC, Racape M, Yoo D, Duong Van Huyen JP, Bruneval P, Taupin JL, Lefaucheur C, Varnous S, Leprince P, Guillemain R, Empana JP, Levine R, Naesens M, Patel JK, Jouven X, Kobashigawa J. Identification and Characterization of Trajectories of Cardiac Allograft Vasculopathy After Heart Transplantation: A Population-Based Study. Circulation. 2020 Jun 16;141(24):1954-1967. doi: 10.1161/CIRCULATIONAHA.119.044924. Epub 2020 May 4. PMID 32363949